CLINICAL TRIAL: NCT06364007
Title: Phase II Study Evaluating the Efficacy of Tremelimumab (T) Plus Durvalumab (D) With Lenvatinib Combined With Concurrent Hepatic Arterial Infusion Chemotherapy (HAIC) in Patients (Pts) With Unresectable Hepatocellular Carcinoma (uHCC)
Brief Title: HAIC Combined With Durvalumab and Tremelimumab and Lenvatinib in uHCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sulai Liu (Other)
Responsible Party: Sponsor-Investigator, Sulai Liu, Hepatobiliary Surgical Department, Hunan Provincial People's Hospital
Organization: Hunan Provincial People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLiu0401
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: HAIC; uHCC; immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treating with a Designed Protocol (Experimental)
  Interventions: Drug: HAIC+STRIDE+Len

INTERVENTIONS:
Drug: HAIC+STRIDE+Len — patients will be administrated with STRIDE plus lenvatinib (8 mg or 12 mg) once daily plus HAIC- modified FOLFOX (oxaliplatin, 85 mg/m2; leucovorin, 400 mg/m2; 5-fluorouracil bolus, 400 mg/m2 on day 1; 5-fluorouracil infusion, 2400 mg/m2 for 46 h).

SUMMARY:
The treatment options for unresectable HCC have rapidly developed, and immunotherapy has shown significant survival benefits in hepatocellular carcinoma. The STRIDE regimen of Single Tremelimumab (high, priming 300-mg dose) Regular Interval Durvalumab (1500 mg every 4 weeks) improved OS vs sorafenib in pts with unresectable HCC. In Asian region, HAIC is applied for HCC patients who are not suitable for surgical resection or local ablation treatment. Retrospective studies suggested a potent antitumor effect and survival benefit of HAIC plus programmed death-1 inhibitor and Lenvatinib. This phase II study was aimed to evaluate the efficacy and safety of STRIDE plus lenvatinib, given concurrently with HAIC in pts with unresectable HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 ~ 70 years old (including 70 years old), male and female;
2. Patients with hepatohcellular carcinoma diagnosed clinically or confirmed by histology / cytology ;
3. Patients with unresectable or metastatic hepatocellular carcinoma;
4. No systematic treatment. Patients recieved previously systematic treatment and progressed can also be included in the group;
5. Patients who underwent hepatectomy in the past should be R0 resection, and the tumor recurrence should be more than 6 months after operation;
6. At least one assessable lesion (mRECIST criteria);
7. Expected survival time ≥ 3 months;
8. ECOG 0 ~ 1;
9. Child Pugh ≤ 7;
10. Be able to cooperate to observe adverse events;
11. Major organs are functioning normally:

    * Hemoglobin ≥ 90 g / L;
    * ANC ≥ 1.5 × 109/L；
    * Platelet count ≥ 75 × 109/L；
    * Albumin ≥ 28 g / L;
    * Total bilirubin ≤ 2 × ULN;
    * AST, ALT ≤ 5 × ULN；
    * ALP ≤ 5 × ULN；
    * Creatinine ≤ 1.5 × ULN；
    * INR or PT ≤ 1.5 × ULN； J) APTT ≤ 1.5 × ULN。

Exclusion Criteria:

1. History of symptomatic congestive heart failure, unstable angina pectoris,
2. Uncontrolled cardia arrhythmia
3. History of hepatic encephalopathy
4. Uncontrolled arterial hypertension
5. Co-infection with HBV and HDV

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
ORR | about 1 year
  objective response rate

SECONDARY OUTCOMES:
PFS | about 1.5 year
  progression-free survival
OS | about 3 year
  overall survival
DCR | about 1 year
  disease control rate
AE | about 3 year
  adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincial People's Hospital(The First Affiliated Hospital of Hunan Normal University), Changsha, Hunan, China